CLINICAL TRIAL: NCT05192707
Title: Standardized Transcutaneous Oxygen Pressure Determination in the Upper Limb: Normal Value and Chronic Limb Ischemia
Brief Title: Transcutaneous Oxygen Pressure (TcPO2) Determination.
Acronym: TcP02
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0545
Record Dates: First submitted 2021-12-02; First posted 2022-01-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Diseases
Keywords: Transcutaneous Oxygen Pressure; Peripheral Arterial Disease; Chronic Limb ischemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Volunteers: TcPO2 measurement in the upper limb of healthy volunteers
  Interventions: Diagnostic Test: TcPO2 measurement on the upper limb
- Patients with arterial disease in the upper limb and wound: Patients with arterial disease in the upper limb and wound (retrospective setting, research on data)
  Interventions: Diagnostic Test: TcPO2 measurement on the upper limb

INTERVENTIONS:
Diagnostic Test: TcPO2 measurement on the upper limb — Measurement of the transcutaneous Oxygen Pressure in the upper limb of 30 healthy volunteers and of at least 30 patients.

SUMMARY:
Upper limb arterial disease is a rare condition compared to lower limb arterial disease. In the lower limb, chronic limb ischemia (CLI) is characterized by an intractable pain or an ulceration present for at least 2 weeks. Guidelines recommend to use Transcutaneous Oxygen pressure (TcPO2) measurement when a CLI is suspected to establish diagnostic with a threshold of 30 mmHg when ankle and toe systolic pressure are not available.

In the upper limb, there is no guideline to define CLI. When there is a wound preventing finger pressure measurement, TcPO2 is theoretically indicated. However, there is neither standardized site to measure nor threshold value of TcPO2.

The investigators hypothesized that normal TcPO2 may be different in the upper limb and that threshold value for CLI may also be different compared to lower limb.

The investigators planned a study with two parts:

1. Prospective study of normal TcPO2 value in healthy volunteers
2. Retrospective analysis of patients with upper limb arterial disease to approach the TcPO2 threshold of CLI allowing healing in upper limb

ELIGIBILITY:
Healthy volunteers part:

Inclusion Criteria:

* healthy volunteer without upper limb arterial disease
* absence of opposition
* affiliated to social insurance

Exclusion Criteria:

* under 18 yrs old
* under law protection
* pregnancy

Retrospective patients part:

Inclusion Criteria:

* patients with a TCPO2 measurement available for the upper limb
* patients with a follow-up of at least 3 months available
* absence of opposition
* affiliated to social insurance

Exclusion Criteria:

* under 18 yrs old
* under law protection
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be made of :
  1. healthy volunteers,
  2. and patients with upper limb arterial disease followed in the "Explorations Fonctionnelles Vasculaires" Unit of the "Médecine Interne" department of Edouard Herriot hospital (HCL, Lyon).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
TcPO2 of the upper limb (blood pressure, measured in millimeters of mercury (mmHg)). | Healthy volunteers: Enrollment. Patients: 1 month after information letter sending.
  Measured on both healthy volunteers (4 sites of measure) and patients with arterial disease The measurements are carried out by non-invasive extracorporeal electrodes with CE (Conformité Européenne) marked equipment and used in accordance with the CE mark.

SECONDARY OUTCOMES:
TcPO2 of the upper limb (mmHg) (only for the healthy volunteers) | Enrollment
  average values of all TcPO2 values.
ROC (Receiving Operator Characteristic) curve for critical ischemia (only for the retrospective patients) | 3 months
  critical ischemia is defined as an amputation more proximal than distal than the electrode or revascularization.
Sensitivity and specificity for critical ischemia (only for the retrospective patients) | 3 months
  critical ischemia is defined as an amputation more proximal than distal than the electrode or revascularization. Tested threshold: 30mmHg, 30 mmHg, 40mmHg, 50mmHg and 60mmHg
patients characteristics (only for the retrospective patients) | 3 months
  age, sex, vascular risk factors, etiology, medical treatment, other treatments).
healing (only for the retrospective patients) | 3 months
  number and percentage of healing without amputation and without revascularization
level of amputation (only for the retrospective patients) | 3 months
  number and percentage of patients with an amputation level more proximal that the electrodes
revascularization (only for the retrospective patient) | 3 months
  number and percentage of revascularization procedures
healing after revascularization | 3 months after revascularization
  percentage of healing following revascularization (only for the retrospective patient if data are available)

CONTACTS AND LOCATIONS:
Overall Officials: Judith CATELLA, MD, Principal Investigator — Service de Médecine Interne - UF Explorations Fonctionnelles Vasculaires, HEH, HCL
Locations (1):
- Service de Médecine Interne - UF Explorations Fonctionnelles Vasculaires, Hôpital Edouard Herriot, Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided